CLINICAL TRIAL: NCT02128139
Title: Infective Endocarditis in Developing Countries, a Prospective, Observational, Multicentre Study
Acronym: EndoDev
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: War Memorial Hospital (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); Oxford University Hospitals NHS Trust (Other); St. Elizabeth Catholic General Hospital Shisong, Cameroun (Unknown); CHU de Brazzaville, Congo Brazzaville (Unknown); Polyclinique International de Bamako, Mali (Unknown); CHR de Saint-Louis Lt Colonel Mamadou Diouf, Sénégal (Unknown); Hôpital Général de Grand Yoff de Dakar, Sénégal (Unknown); Bafoussam Regional Hospital, Cameroon (Unknown); Hospital Laquinitinie de Douala (Unknown); Yaounde Central Hospital (Other Government); National Hospital of Niamey (Other); Centre National Hospitalier Universitaire de Pneumo-Phtisiologie de Cotonou, Benin (Unknown); Hospital General De Douala (Other); Eduardo Mondlane University (Other); Laos Oxford Mahosot Wellcome Research Unit (Unknown); Mulago Hospital, Uganda (Other); Fann Hospital, Senegal (Unknown); Institute of Cardiology Abidjan (Unknown)
Responsible Party: Sponsor
Other Study IDs: C12-37 / EndoDev; Cardiology and Development (Other: INSERM)
Record Dates: First submitted 2013-12-17; First posted 2014-05-01 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Infective Endocarditis
Keywords: Infective endocarditis; Developing country; Global health; Cardiac surgery; Heart valve disease; Bacteremia
MeSH Terms: conditions — Endocarditis; Heart Valve Diseases; Bacteremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Introduction. Comprehensive data on infective endocarditis in developing countries are scarce.

Objectives: Description of the characteristics (clinical and microbiological) and assessment of the outcomes of infective endocarditis in low-income countries.

Methods : Prospective, Observational, Multicentre study. Inclusion criteria: patients aged over 1 year fulfilling the modified Duke criteria for infective endocarditis.

Exclusion criteria: patient included during a previous infective endocarditis episode.

Outcomes measures: Mortality at 6 months follow-up; mortality at 1 month follow-up; access to antibiotic treatment (modalities and duration), hospital length of stay and reason for discharge, and cardiac surgery when indicated.

Duration: One year (June 2014- June 2015)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 1 year diagnosed with infective endocarditis according to the modified Duke criteria

Exclusion Criteria:

* Already included for a previous episode of infective endocarditis (i.e., relapse or reinfection)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital-based population.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Mortality at 1 month follow-up | 1 month

SECONDARY OUTCOMES:
Mortality at 6 months follow-up | 6 months

OTHER OUTCOMES:
Access to cardiac surgery | 6 months
  Heart surgery is not available in many low-income countries. One of the objectives is to assess whether guidelines can be applied in low-secourced settings.

CONTACTS AND LOCATIONS:
Locations (6):
- Joseph Kado, Suva, Fiji
- Paul N. Newton, Vientiane, Laos
- Beatriz Ferreira, Maputo, Mozambique
- Senegal (2):
  - Abdul Kane, Dakar
  - Bara Diop, Dakar
- Emmy Okello, Kampala, Uganda